CLINICAL TRIAL: NCT01065779
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of FOSAMAX PLUS and FOSAMAX PLUS D in Usual Practice
Brief Title: FOSAMAX PLUS and FOSAMAX PLUS D Re-examination Study (0217A-267)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0217A-267; 2010_007
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Fumigant 93

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOSAMAX PLUS or FOSAMAX PLUS D: Patients with Osteoporosis treated with FOSAMAX PLUS (70 mg/2800 IU) or FOSAMAX PLUS D (70 mg/5600 IU).
  Interventions: Drug: FOSAMAX PLUS; Drug: FOSAMAX PLUS D

INTERVENTIONS:
Drug: FOSAMAX PLUS — Patients with Osteoporosis treated with FOSAMAX PLUS (70 mg alendronate/2800 International Units (IU) Vitamin D). One tablet taken once weekly.
Drug: FOSAMAX PLUS D — Patients with Osteoporosis treated with FOSAMAX PLUS D (70 mg alendronate/5600 IU Vitamin D). One tablet taken once weekly.

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of FOSAMAX PLUS / FOSAMAX PLUS D through collecting the safety information according to the Re-examination Regulation for New Drugs.

Note: FOSAMAX PLUS D is known as FOSAMAX PLUS in several markets. FOSAMAX PLUS (70 mg/2800 IU) and FOSAMAX PLUS D (70 mg/5600 IU).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are treated with FOSAMAX PLUS / FOSAMAX PLUS D within label for the first time

Exclusion Criteria:

* Participants who have a contraindication to FOSAMAX PLUS / FOSAMAX PLUS D according to the current local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Osteoporosis treated with FOSAMAX PLUS or FOSAMAX PLUS D
Sampling Method: Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- FOSAMAX PLUS/ FOSAMAX PLUS D: Participants with Osteoporosis treated with FOSAMAX PLUS or FOSAMAX PLUS D. One 70 mg alendronate/2800 International Units (IU) Vitamin D tablet or one 70 mg alendronate/5600 IU Vitamin D tablet taken once weekly.
Period: Overall Study
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Started | 880
Completed | 798
Not Completed | 82
Not completed — Duplicate Investigation | 1
Not completed — Investigation Before Contract Date | 37
Not completed — Non-enrollment Period Administration | 10
Not completed — Not Administered With Study Drug | 17
Not completed — Failed to Follow-up | 10
Not completed — Inclusion Criteria Violation | 7

BASELINE CHARACTERISTICS:
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 880
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.12 (9.05)
Sex/Gender, Customized [Number; unit: participants]
  Female | 741
  Male | 57
  Excluded from Analysis | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants that experienced Serious Adverse events (SAE). There was no required routine visit scheduled for AE assessment. AEs were collected through participant self-reporting and assessed by investigators.
  SAEs were considered serious if the event resulted in:
  * death or was life-threatening
  * prolonged an existing inpatient hospitalization
  * a persistent or significant disability/ incapacity
  * a congenital anomaly/ birth defect
  * a significant medical situation, other important medical event based upon appropriate medical judgment of the investigator
Time Frame: Up to ~ 16 weeks and 14 days after treatment discontinuation
Population: Safety evaluation was performed in participants who took at least one dose of study medication and completed > 1 follow up visit.
Measure: Number; unit: Participants
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 798
Participants | 0

2. Primary Outcome: Number of Participants With Unexpected Adverse Events
Description: Number of participants that experienced unexpected Adverse Events (AEs) regardless of whether or not the AE was considered related to the use of the product. There was no required routine visit scheduled for AE assessment. An AE was defined as any unfavorable & unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product. Any worsening (any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also considered an AE.
Time Frame: Up to ~ 16 weeks and 14 days after treatment discontinuation
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 798
Participants | 2

3. Primary Outcome: Number of Participants With Non-Serious AEs
Description: An AE was defined as any unfavorable & unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the product, was also considered an AE. There was no required routine visit scheduled for AE assessment. AEs were collected through participant self-reporting and assessed by investigators.
Time Frame: Up to ~ 16 weeks and 14 days after treatment discontinuation
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 798
Participants | 42

4. Primary Outcome: Number of Participants With Improved, Unchanged, or Worsened Disease
Description: Evaluation of disease improvement was conducted in 3 categories of "improved", "unchanged", or "worsened". Changes in biochemical markers and vitamin D levels were reviewed before (baseline) and after treatment using statistical analyses to determine disease status, which was reported as either "improved", "unchanged", or "worsened".
Time Frame: Baseline and end of Treatment (Up to ~ 16 weeks)
Population: Among 798 participants in safety evaluation, there was a total of 789 participants for efficacy evaluation excluding 8 participants who took study drug for < 4 weeks and 1 participant who did not enter efficacy evaluation.
Measure: Number; unit: Participants
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 789
Participants
  Improved | 549
  Unchanged | 239
  Worsened | 1

5. Primary Outcome: Change From Baseline in Serum 25-hydroxyvitamin D at End of Treatment
Description: For efficacy evaluation, changes in Serum 25-hydroxyvitamin D were evaluated before study drug administration and at end of study drug treatment. Change was calculated as the later time point (at ~16 weeks) minus the earlier time point (baseline). The Last Observation Carried Forward (LOCF) method was used. That is, the last observed non-missing value was used to fill in missing values at the later point in the study.
Time Frame: Baseline and End of Treatment (Up to ~ 16 weeks)
Population: Among 798 participants in safety evaluation, there was a total of 789 participants for efficacy evaluation excluding 8 participants who took study drug for < 4 weeks and 1 participant who did not enter efficacy evaluation. Only participants with lab values submitted to Sponsor were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 10
ng/mL | 1.73 (1.48)

6. Primary Outcome: Change From Baseline in Serum Osteocalcin at End of Treatment
Description: For efficacy evaluation, changes in Serum Osteocalcin were evaluated before study drug administration and at end of study drug treatment. Change was calculated as the later time point (at ~16 weeks) minus the earlier time point (baseline). The Last Observation Carried Forward (LOCF) method was used. That is, the last observed non-missing value was used to fill in missing values at the later point in the study.
Time Frame: Baseline and End of Treatment (Up to ~ 16 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 10
ng/mL | 0.69 (0.32)

7. Primary Outcome: Change From Baseline in Urine Deoxypyridinoline at End of Treatment
Description: For efficacy evaluation, changes in Serum Deoxypyridinoline were evaluated before study drug administration and at end of study drug treatment. Change was calculated as the later time point (at ~16 weeks) minus the earlier time point (baseline). The Last Observation Carried Forward (LOCF) method was used. That is, the last observed non-missing value was used to fill in missing values at the later point in the study.
Time Frame: Baseline and End of Treatment (Up to ~ 16 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nmol/mmol
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 11
nmol/mmol | 1.03 (0.83)

8. Primary Outcome: Change From Baseline in Alkaline Phosphatase at End of Treatment
Description: For efficacy evaluation, changes in Serum Alkaline Phosphatase were evaluated before study drug administration and at end of study drug treatment. Change was calculated as the later time point (at ~16 weeks) minus the earlier time point (baseline). The Last Observation Carried Forward (LOCF) method was used. That is, the last observed non-missing value was used to fill in missing values at the later point in the study.
Time Frame: Baseline and End of Treatment (Up to ~ 16 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Number analyzed (Participants) | 33
mg/dL | -16.36 (37.58)

ADVERSE EVENTS:
Time Frame: Up to ~ 16 weeks and 14 days after treatment discontinuation.
Description: Safety evaluation was performed in participants who took at least one dose of study medication and completed > 1 follow up visit.
Arm/Group | FOSAMAX PLUS/ FOSAMAX PLUS D
Serious Adverse Events (participants affected / at risk) | 0/798
Other Adverse Events (participants affected / at risk) | 0/798

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No